CLINICAL TRIAL: NCT00252382
Title: Phase 2 Open-Label, Multicenter Clinical Study of the Safety and Efficacy of the Intravenous Administration of SNS-595 as Second-Line Chemotherapy in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Efficacy Clinical Study of SNS-595 for Second-Line Therapy in Patients With Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0005
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2017-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung; Squamous Cell; Large Cell; Adenocarcinoma; Carcinoma; Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Carcinoma; Neoplasms | interventions — vosaroxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Treatment with 48 mg/m2 of SNS-595 (Experimental): Patients are treated with 48 mg/m2 of the drug SNS-595 injection once every 21 days for up to 6 cycles as a second -line therapy to patients with advanced non-small cell lung cancer (NSCLC)
  Interventions: Drug: SNS-595 Injection

INTERVENTIONS:
Drug: SNS-595 Injection — Vosaroxin (formerly voreloxin or SNS-595) is a first in class anticancer quinolone derivative, non anthracycline topoisomerase II inhibitor. It induces replication dependent DNA damage by intercalating DNA and inhibiting topoisomerase II, leading to apoptosis.
  Other Names: Voreloxin; Vosaroxin

SUMMARY:
The purpose of this study is to evaluate the objective tumor response rate (based on the RECIST criteria) to SNS-595 as a second-line therapy in patients with advanced NSCLC.

DETAILED DESCRIPTION:
Other objectives of this study are to assess the safety, tumor response, time to disease progression, survival rate and to explore several potential biomarkers to see how these levels change after administration of SNS-595.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign a written informed consent document
* Patients who have recurrent or metastatic NSCLC, who have failed initial therapy with a platinum-containing regimen and have not received any second-line therapy (adjuvant therapy is acceptable if it was completed greater than or equal to 12 months before the cancer recurrence)
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Laboratory Values within the normal or reasonable reference range as specified by the protocol

Exclusion Criteria:

* Prior exposure to SNS-595
* Pregnant or breastfeeding
* Women of childbearing potential or male partners of women of childbearing potential unwilling to use an approved, effective means of contraception according to the institution's standards
* Other active malignancies or other malignancies within the past 12 months except non-melanoma skin cancer, cervical intraepithelial neoplasia or prostatic intraepithelial neoplasia
* Brain metastases, if present, without radiologic evidence of progressive disease for at least 3 months after completion of therapy
* Myocardial infarction, cerebrovascular accident/transient ischemic attack (TIA) or thromboembolic event (deep vein thrombosis or pulmonary embolus) within 6 months before the first SNS-595 dose
* Requires kidney dialysis (hemodialysis or peritoneal)
* Prior chemotherapy, investigational agents, or radiation therapy within 28 days before Cycle 1 Day 0; however, nitrosoureas and mitomycin are not permitted for at least 42 days before Cycle 1 Day 0
* In patients with toxicities caused by prior cancer therapy, those toxicities must have returned to less than or equal to Grade 1, with the exception of alopecia
* Prior pelvic radiation therapy or radiation to greater than or equal to 25% of bone marrow reserve (prior palliative radiation is permitted as long as it does not exceed 25% of bone marrow reserve)
* Any other medical, psychological, or social condition that, in the opinion of the Principal Investigator, would contraindicate the patient's participation in the clinical trial due to safety concerns or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-12-27 (Actual); Primary Completion 2007-03-05 (Actual); Study Completion 2007-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Michelson, MD, Study Director — Sunesis Pharmaceuticals
Locations (4):
- United States (4):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Duke Comprehensive Cancer Center, Duke University, Durham, North Carolina
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With 48 mg/m2 of SNS-595
Started | 31
Completed | 5
Not Completed | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Open label administration of SNS-595 48 mg/m2 treatment on day one of 21 day cycles, up to 6 cycles.
Arm/Group | Total
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participant at entry.
  years | 60.4 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate
Description: ORR is based on RECIST criteria to SNS-595 as a second-line therapy in patients with advanced NSCLC. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 168 days
Population: Efficacy Analysis Population
Measure: Count of Participants; unit: Participants
Groups:
- Total: SNS-595 48 mg/m2
Arm/Group | Total
Number analyzed (Participants) | 26
Participants | 1

2. Secondary Outcome: Best Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions; >=20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions (PD); Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (SD). The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started).
Time Frame: 168 days
Population: Efficacy Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Total
Number analyzed (Participants) | 26
Participants
  Partial Response | 1
  Progressive Disease | 17
  Stable Disease | 8

ADVERSE EVENTS:
Time Frame: 196 days
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 14/31
Serious Adverse Events (participants affected / at risk) | 6/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia pneumococcal (Infections and infestations) | 1
Depression (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=31)
Anaemia (Blood and lymphatic system disorders) | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal tenderness (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Hiatus hernia (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Lip disorder (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 17
Oesophagitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal spasm (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Disease progression (General disorders) | 1
Fatigue (General disorders) | 21
Non-cardiac chest pain (General disorders) | 4
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Fungal infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Breath sounds abnormal (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to bone (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Coordination abnormal (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Sensory loss (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Micturition disorder (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Night sweats (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Nasal sinus drainage (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Statistical fields are not included here because no statistical testings were performed to compare any treatment group. No p-values or odds ratios were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days